CLINICAL TRIAL: NCT05282953
Title: A Phase I/II Dose-escalating Study of the Safety, Tolerability and Efficacy of KIO-301 Administered Intravitreally to Patients With Retinitis Pigmentosa and Choroideremia (ABACUS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kiora Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIO-301-1101
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Retinitis Pigmentosa; Choroideremia; Non-Syndromic Rod-Dominant Inherited Retinal Diseases
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Retinitis Pigmentosa and Choroideremia (Experimental)
  Interventions: Drug: KIO-301

INTERVENTIONS:
Drug: KIO-301 — KIO-301 intravitreal injection at ascending doses

SUMMARY:
A phase I/II dose-escalating study of the safety, tolerability and efficacy of KIO-301 administered intravitreally to patients with retinitis pigmentosa and choroideremia (ABACUS).

DETAILED DESCRIPTION:
Main Study: assesses the safety and tolerability of single doses of KIO-301 when administered intravitreally to participants with retinitis pigmentosa and choroideremia.

Sub-study: determines the test/re-test reliability of functional vision assessments in participants with low visual acuity.

ELIGIBILITY:
Main Study:

Inclusion Criteria

1. Be aged 18 to 80 years at Visit 1 of either sex and of any race.
2. Be willing and able to provide informed consent either written, or if the Participant is not able to read, provide consent as stipulated by local laws and Human Research Ethics Committee (HREC) guidelines.
3. Be willing and able to follow all instructions and attend all study visits.
4. Have a clinical diagnosis of retinitis pigmentosa (Cohorts 1 - 3) or choroideremia (Cohort 3 only).
5. Have a visual acuity of:

   1. no light perception for Cohort 3 or
   2. no light perception or bare light perception for Cohort 1 confirmed with a LogMar > 2.9 using the Berkeley Rudimentary Vision Test (BRVT), or
   3. count fingers or hand motion for Cohort 2 as confirmed by a LogMar ≤ 2.9 and > 1.6 using the BRVT.
6. Have similar visual acuity in both eyes as defined as a LogMar difference between eyes of < 0.05 using the BRVT.
7. Be willing to avoid disallowed medications and treatments for the duration of the study.
8. Contraception:

   * If female, agree to submit to a pregnancy test at Visit 1, or not be of childbearing potential. All participants of childbearing potential must agree to use an acceptable method of contraception for the duration of the study. Acceptable methods of birth control include oral, transdermal, injectable, or implantable contraception, intrauterine device, abstinence, and surgical sterilisation of partner. Female Participants are not of childbearing potential if they have had a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or are post-menopausal by at least 12 months.
   * Male participants will be surgically sterile for at least 3 months, or when sexually active with female partners of childbearing potential will be required to use a male condom from Screening until 3 months the last dose of study drug. Sexual intercourse with female partners who are pregnant, or breastfeeding should be avoided unless condoms (or double barrier method) are used from the time of the first dose until 3 months after the last dose of study drug. Male participants are required to refrain from donation of sperm from Screening until 3 months after the last dose of study drug.
   * Participants who have practiced true abstinence for at least 1 year because of the participant's lifestyle choice (i.e., the participant should not become abstinent just for the purpose of study participation) are exempt from contraceptive requirements. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. If a participant who is abstinent at the time of signing the ICF becomes sexually active they must agree to use contraception as described above and as outlined in the ICF.
   * For participants who are exclusively in same sex relationships, contraceptive requirements do not apply. If a participant who is in a same sex relationship at the time of signing the ICF becomes engaged in a heterosexual relationship, they must agree to use contraception as described above and as outlined in the ICF.

Exclusion Criteria

1. Have evidence of material/substantial optic nerve disease.
2. Have a history of retinal detachments.
3. Have clinically significant ocular disease (e.g., corneal oedema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study or clinically significant opacities of the media.
4. Have high intraocular pressure (IOP) >22 mm Hg.
5. Have had a previous intraocular surgery (excluding phakocataract surgery).
6. Have aphakia.
7. Have a psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to Screening, a history of suicide plan.
8. Have any clinically significant abnormality at Screening determined by medical history, vital signs, blood chemistry, haematology, urinalysis or a 12-lead electrocardiogram (ECG), as assessed by the investigator.
9. Have any other medical condition or significant co-morbidities, or any finding during Screening, which in the view of the Investigator is likely to interfere with the study or put the Participant at risk, confound study data, or interfere significantly with study participation.
10. Have clinical signs of active infection and/or a temperature greater than 38.0°C at the time of Screening. Study entry may be deferred at the discretion of the Principal Investigator (PI).
11. Have implanted pacemakers.
12. Have intracranial aneurysm clips.
13. Have cochlear implants.
14. Have implanted drug infusion and prosthetic devices.
15. Have certain intrauterine contraceptive devices.
16. Have any other type of metal implant or object such as shrapnel, pins, screws or wire mesh.

Sub-study:

Inclusion Criteria

1. Patients with RP, CHM, or other non-syndromic, rod-dominant IRDs, and a visual acuity of:

   1. NLP OU confirmed by inability to see pen torch light at 25cm in OD, OS, and OU (assigned logMAR of 4.0 as per BRVT).
   2. Light perception (LP), Ultra Low Vision (ULV), or Low Vision (LV) OU (logMAR > 1.0 and < 4.0) as determined by the BRVT or Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.
2. Aged 18 years or older and of either sex and of any race.
3. Willing and able to provide informed consent either written, or if the Participant is not able to read, provide consent as stipulated by local laws and HREC guidelines.
4. Willing and able to attend all study visits and perform study assessments.

Exclusion Criteria

1. Have any evidence of any other material/substantial disease that, in the opinion of the investigator, is likely to interfere with the study objectives or put the Participant at risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Main Study Primary Outcome Measure | 84 days.
  Number of participants with treatment-related adverse events as assessed by overall changes in retinal thickness and appearance, clinical chemistry and hematology, and other eye assessments.

OTHER OUTCOMES:
Sub-study Outcome Measure | 42 days.
  Test/re-test reliability of functional vision assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Casson, Principal Investigator — Royal Adelaide Hospital
Locations (3):
- Australia (3):
  - Save Sight Institute, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Harley Eye Clinic, North Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No